CLINICAL TRIAL: NCT03705585
Title: CVD 38000: Immunity, Microbiome, Epigenetics, and a Systems Biology Approach to the Study of Responses to Vaccination With Typhoid and/or Cholera
Brief Title: CVD 38000: Study of Responses to Vaccination With Typhoid and/or Cholera
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Bruce Greenwald, Professor of Medicine, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00081568
Record Dates: First submitted 2018-10-04; First posted 2018-10-15 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Typhoid and/or Cholera Vaccination
MeSH Terms: interventions — Vaxchora; cholera vaccine CVD 103-HgR

STUDY DESIGN:
Intervention Model Description: Volunteers who choose to take part in this study will receive the licensed FDA approved Oral Typhoid Vaccine (Vivotif) and/or the licensed FDA approved Oral Cholera Vaccine (Vaxchora). Volunteers also have the possibility of being a control participant who will not be vaccinated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Vaccination, Endoscopy (Experimental): Individuals receive immunization with Vivotif typhoid vaccine and/or Vaxchora cholera vaccine prior to routine endoscopic examination. During endoscopy, small bowel biopsies will be obtained to examine immune responses and microbiota at the mucosal level; brushings might also be obtained.
  Interventions: Drug: Vivotif Typhoid Oral Vaccine; Drug: Vaxchora
- Endoscopy, Vaccination, Endoscopy (Experimental): Individuals receive immunization with Vivotif typhoid vaccine and/or Vaxchora cholera vaccine after initial endoscopic exam and specimen collection and prior to a routine follow up endoscopic examination during which additional specimens will be collected.
  Interventions: Drug: Vivotif Typhoid Oral Vaccine; Drug: Vaxchora
- Endoscopy Without Vaccination (No Intervention): Individuals do not receive immunization but consent to collection of specimens during endoscopy. The specimens to be collected in all three groups include stool, saliva, and small bowel biopsies (terminal ileum if colonoscopy performed, duodenum if EGD performed).

INTERVENTIONS:
Drug: Vivotif Typhoid Oral Vaccine — The 4 doses (1 capsule each) will be administered on alternate days, e.g., days 0, 2, 4, and 7 (± 1 day) under the supervision of the study coordinator(s).
  Other Names: Ty21a Typhoid Oral Vaccine
  Arms: Endoscopy, Vaccination, Endoscopy; Vaccination, Endoscopy
Drug: Vaxchora — One dose. Approximately 100 mL of cool or room temperature purified bottled water is placed into a clean disposable cup. The contents of the buffer sachet are added to the water and stirred. Then the contents of the active (lyophilized vaccine) sachet are added to the water and stirred for approximately 30 seconds. The reconstituted mixture should be completely ingested within 15 minutes.
  Other Names: CVD 103-HgR
  Arms: Endoscopy, Vaccination, Endoscopy; Vaccination, Endoscopy

SUMMARY:
This is an open-label, non-randomized study. The purpose of this study is to better understand how vaccines against typhoid fever and cholera affect the normal immune system and bacteria in the intestine. Patients having standard-of-care endoscopies (colonoscopy and/or esophagogastroduodenoscopy (EGD)) will be divided into 3 groups:

Group 1: Vivotif typhoid vaccination and/or Vaxchora cholera vaccination then endoscopy Group 2: Endoscopy, then Vivotif typhoid vaccination and/or Vaxchora cholera vaccination, then follow-up endoscopy Group 3: Endoscopy without vaccination.

Both vaccines used in this study are licensed by the Food and Drug Administration (FDA) for travelers to developing countries. Volunteers will be asked to donate tissue, blood, saliva and stool samples for studying how the body responds to the typhoid and/or cholera vaccine.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 years and older
* 2. Already scheduled to undergo an EGD or colonoscopy for screening, surveillance, or a medically-indicated work-up at the University of Maryland Medical Center (main campus or Midtown)
* 3. Able to provide written informed consent prior to initiation of any study procedures
* 4. Healthy, as defined by considered fit to undergo outpatient elective EGD/colonoscopy by the evaluating health care provider

Exclusion Criteria:

* 1. Pregnancy or nursing mother
* 2. Known coagulopathy or bleeding disorder preventing mucosal biopsy
* 3. History of Crohn's disease or ulcerative colitis
* 4. For Subjects undergoing lower endoscopy (colonoscopy) only: Surgical removal of the ileocecal valve or any part of the small or large intestine (non-complicated appendectomy will be considered eligible)
* 5. Allergic reaction to oral typhoid or cholera vaccine in the past
* 6. Immunosuppression from illness or treatment, including

  1. immune-deficiency disorders such as Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS)
  2. leukemia, lymphoma, or cancers (localized non-melanoma skin cancers which are deemed inactive should be considered eligible)
* 7. Receipt of any other vaccine two weeks prior to receipt of Ty21a or CVD 103-HgR
* 8. Positive urine pregnancy test (HCG) prior to colonoscopy or vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Responders | approximately 5 years
  Percentage of responders by cytokine production (Interferon-gamma (IFN-gamma) or Tumor Necrosis Factor-alpha (TNF-α)) by mass cytometry or flow cytometry. Responders will be defined as those volunteers showing increases post-immunization of >0.1% of positive CD8+ cells for IFN-gamma or TNF-α over baseline (pre-immunization) values.) or Tumor Necrosis Factor-alpha (TNF-α)) by mass cytometry or flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No